CLINICAL TRIAL: NCT04937582
Title: Long Term Cognitive and Psychological Disorders After Severe COVID-19 Infection in Young Patients
Brief Title: Cognitive and Psychological Disorders After Severe COVID-19 Infection
Acronym: NEUROCOG-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Régional Metz-Thionville (Other); Centre hospitalier Epinal (Unknown); Hopitaux Civils de Colmar (Other)
Responsible Party: Principal Investigator, Lucie HOPES, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00447-34
Record Dates: First submitted 2021-05-28; First posted 2021-06-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: COVID 19
Keywords: COVID 19 cognitive impairement
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Confirmed cognitive disorder (Experimental): Patients with abnormal QPC score at screening visit and confirmed cognitive disorder on the neuropsychological assessment during Visit V1.
  Intervention Completed by MRI (magnetic resonance imaging), EEG (Electroencephalogram) and possible psychiatric evaluation at Visit 1B.
  Follow-up 2 years after initial hospitalisation (Visit 2 : neuropsychological assessment ; if needed MRI, EEG, lumbar puncture)
  Interventions: Diagnostic Test: Cognitive assessment; Diagnostic Test: Imaging; Diagnostic Test: Routine care; Other: Psychiatric evaluation
- Absence of cognitive disorder (Experimental): Patients with abnormal QPC score at screening and absence of cognitive disorder on the neuropsychological assessment during Visit V1.
  Interventions: Diagnostic Test: Cognitive assessment; Other: Psychiatric evaluation

INTERVENTIONS:
Diagnostic Test: Cognitive assessment — Complete cognitive and psychological assessment
Diagnostic Test: Imaging — Brain MRI
  Optional: Brain FDG PET (Brain positron emission tomography with F-18 fluorodeoxyglucose)
  Arms: Confirmed cognitive disorder
Diagnostic Test: Routine care — Electroencephalogram (EEG)
  Optional: polysomnography, lumbar puncture
  Arms: Confirmed cognitive disorder
Other: Psychiatric evaluation — Psychiatric consultation if necessary
  Arms: Confirmed cognitive disorder
Other: Psychiatric evaluation — Psychiatric consultation if necessary (before the end of their participation in the study)
  Arms: Absence of cognitive disorder

SUMMARY:
As COVID-19 pandemic is still ongoing, patients follow-up begins to reveal cognitive and psychological disorders. There are not yet well described, neither their physiopathology. This study will consist in the detection and characterization of cognitive and psychological impairments in young patients under 65 years of age who have been hospitalized more than 72 hours for a severe COVID-19 infection.

DETAILED DESCRIPTION:
Initial consecutive screening of patients (<65 years) hospitalized between the 01/10/2020 and the 01/07/2021 for more than 72 hours for COVID-19 infection in 6 hospitals of the East of France. If detection of cognitive complaints (QPC scale : Questionnaire of cognitive complaints), continuation of the study.

Evaluation with cognitive assessments, morphological and functional imaging and EEG will be done at 9 ± 3 months and 2 years after initial hospitalisation. Data will be collected concerning social and professional outcome.

An ancillary study will be conducted at the Nancy University Hospital. This ancillary study is entitled "TRAUMA-COV: Screening and therapeutic proposal of post-traumatic sequelae in the aftermath of a severe Covid-19 in young subjects". The main objective of this study is to evaluate the incidence of post-Covid-19 post-traumatic disorders (post-traumatic stress disorder, psychogenic and somatoform dissociative tendency, neurological dissociative disorder) in a longitudinal way. This optional study will be offered to all patients from the main study who meet the selection criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age (at discharge of hospitalization),
* Patient hospitalized for more than 72 hours (in intensive care or conventional sector) for a COVID-19 infection defined by a positive PCR (Polymerase Chain Reaction) test and/or typical aspect on thoracic scanner,
* Patient discharged from hospital between 01/10/2020 and 01/04/2021,
* Patient with suspected cognitive impairment (obtaining a pathologic QPC score) during the phone screening,
* Patient having received complete information on the organization of the research and having given written informed consent (or a third person, independent of the investigator and the sponsor, in case of inability to read or write),
* Patient affiliated with a social security plan or beneficiary of such a plan,
* Patient with a sufficient level of written French comprehension to complete the cognitive assessment.

Exclusion Criteria:

* Inability to travel to perform the BNP or additional tests,
* Contraindication to perform brain MRI (pacemaker, etc.),
* Presence of chronic neurological diseases (multiple sclerosis, neurodegenerative disease, epilepsy) and/or major cognitive disorders (stroke, head trauma) pre-COVID-19,
* Presence of psychiatric disorder historys (bipolar or psychotic illness) pre-COVID-19,
* Patients with very extensive post-COVID-19 brain damage leading to impossibility to realise cognitive assessment,
* Addictive history or comorbidities (alcoholism, drug use) with sequelae of cognitive impairment,
* Persons covered by articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Characterization of cognitive and psychological disorders 1 year after COVID-19 infection | up to 1 year
  Perfomance to cognitive assessment

SECONDARY OUTCOMES:
Frequency of cognitive and psychological disorders 1 year and 2 years after COVID-19 infection | up to 2 years
  Number of patients with confirmed cognitive and/or psychological disorder compared to the total number of patients who completed the QPC scale
Severity of cognitive and psychological disorders 1 year after COVID-19 infection | up to 1 year
  Perfomance to cognitive assessment
Evaluate the prognosis of cognitive and psychological disorders at 2 years according to the proposed medical care | up to 2 years
  Cognitive assessment
Evaluate the prognosis of cognitive and psychological disorders at 2 years according to the proposed medical care | up to 2 years
  Change from baseline in professional status

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Department of Neurology, Nancy, France

IPD SHARING:
Plan to Share IPD: No